CLINICAL TRIAL: NCT01181349
Title: Incidence of Postoperative Residual Neuromuscular Blockade - A Multicenter, Observational Study in Portugal
Brief Title: Incidence of Incomplete Postoperative Neuromuscular Recovery From Anesthesia (P07535)(Completed)
Acronym: INSPIRE
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P07535
Record Dates: First submitted 2010-07-23; First posted 2010-08-13 (Estimated); Results first posted 2012-04-02 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Neuromuscular Blockade
Keywords: neuromuscular blockade; general anesthesia
MeSH Terms: interventions — Neuromuscular Blocking Agents

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- P07535 study participants with a TOF ratio <0.9: Participants enrolled in the P07535 study who are included in the primary outcome measurement, which is defined as the incidence of postoperative residual neuromuscular blockade, who had a TOF ratio <0.9 at PACU arrival.
  Interventions: Other: Neuromuscular Blocking Agent (NMBA)
- P07535 study participants with a TOF ratio ≥0.9: Participants enrolled in the P07535 study who are included in the primary outcome measurement, which is defined as the incidence of postoperative residual neuromuscular blockade, who had a TOF ratio ≥0.9 at PACU arrival.
  Interventions: Other: Neuromuscular Blocking Agent (NMBA)

INTERVENTIONS:
Other: Neuromuscular Blocking Agent (NMBA) — While neuromuscular blockade drug(s) are involved in this study prior to actual study initiation (this is an observational study), it should be noted that the identity, combination(s), and dosages of these drugs (also referred to as general anesthesia drug[s]) are not specified in the protocol.
  Groups: P07535 study participants with a TOF ratio <0.9
Other: Neuromuscular Blocking Agent (NMBA) — While neuromuscular blockade drug(s) are involved in this study prior to actual study initiation (this is an observational study), it should be noted that the identity, combination(s), and dosages of these drugs (also referred to as general anesthesia drug[s]) are not specified in the protocol.
  Groups: P07535 study participants with a TOF ratio ≥0.9

SUMMARY:
This is a multicenter, observational study in adult participants undergoing different types of elective surgical procedures requiring general anesthesia. During the first study period, there will be a cross-sectional evaluation of neuromuscular blockade level upon participant arrival at Post Anesthesia Care Units (PACUs). During the second study period, hospital discharge data from the participants will be collected. The purpose of this study is to determine the incidence of incomplete postoperative neuromuscular recovery from anesthesia at PACUs in Portuguese hospitals. This is a cross-sectional and retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Informed consent signed
* Admission for elective surgery
* Administration of nondepolarizing NMBAs during surgery

Exclusion Criteria:

* Admission for emergency surgery
* Reoperation on the same hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Portuguese participants undergoing different types of elective surgical procedures requiring general anesthesia with neuromuscular blocking agents
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

REFERENCES:
- [Derived] Esteves S, Martins M, Barros F, Barros F, Canas M, Vitor P, Seabra M, Castro MM, Bastardo I. Incidence of postoperative residual neuromuscular blockade in the postanaesthesia care unit: an observational multicentre study in Portugal. Eur J Anaesthesiol. 2013 May;30(5):243-9. doi: 10.1097/EJA.0b013e32835dccd7. PMID 23344123

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Adult study participants undergoing different types of elective surgical procedures requiring general anesthesia
  with neuromuscular blocking agents
Period: Overall Study
Arm/Group | All Participants
Started | 350
Completed | 350
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216
  Male | 134

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Train-of-four (TOF) Ratio <0.9 at PACU Arrival
Description: The incidence of incomplete postoperative neuromuscular recovery from general anesthesia was assessed in study participants upon arrival in the PACU, after their respective surgical procedures were completed. Neuromuscular functioning was assessed by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. The TOF ratio is the ratio of the magnitude of the fourth twitch to that of the first twitch, and a ratio <0.9 indicates residual neuromuscular blockade (incomplete neuromuscular recovery).
Time Frame: Upon arrival in the PACU
Population: Full analysis set (FAS) population includes all treated participants
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 350
participants | 91

2. Secondary Outcome: Number of Participants With and Without Postoperative Residual Neuromuscular Blockade Who Received Identified Neuromuscular Blocking Agents
Description: Neuromuscular blocking agents administered to participants undergoing surgical procedures were recorded. The number of participants who received atracurium, cisatracurium, rocuronium or vecuronium is presented, for participants with and without residual neuromuscular blockade.
Time Frame: From start of surgery through PACU arrival
Population: FAS population includes all treated participants; for this outcome measure only participants who received atracurium, cisatracurium, rocuronium or vecuronium are included
Measure: Number; unit: participants
Groups:
- P07535 Study Participants With a TOF Ratio <0.9: Participants with TOF ratio <0.9 upon arrival at PACU, defined as indicating presence of residual neuromuscular blockade
- P07535 Study Participants With a TOF Ratio ≥0.9: Participants with TOF ratio ≥0.9 upon arrival at PACU, defined as indicating absence of residual neuromuscular blockade
Arm/Group | P07535 Study Participants With a TOF Ratio <0.9 | P07535 Study Participants With a TOF Ratio ≥0.9
Number analyzed (Participants) | 87 | 250
participants
  Participants Receiving Atracurium | 13 | 42
  Participants Receiving Cisatracurium | 35 | 73
  Participants Receiving Rocuronium | 31 | 118
  Participants Receiving Vecuronium | 8 | 17
Statistical Analysis 1: Comparison: P07535 Study Participants With a TOF Ratio <0.9 vs P07535 Study Participants With a TOF Ratio ≥0.9; Cross tables were performed between TOF ratio and medications administered. Statistical significance was evaluated using Chi-square test or Fisher's Exact Test. All tests were performed at a significance level of 0.05; Test type: Superiority or Other; p = 0.169, Chi-square test or Fisher's Exact Test

3. Secondary Outcome: Number of Participants With and Without Postoperative Residual Neuromuscular Blockade Who Received Propofol or Sevoflurane
Description: Anesthetic agents administered to participants undergoing surgical procedures were recorded. The number of participants who received propofol or sevoflurane is presented, for participants with and without residual neuromuscular blockade.
Time Frame: From start of surgery through PACU arrival
Population: FAS population includes all treated participants; for this outcome measure only participants who received propofol or sevoflurane are included
Measure: Number; unit: participants
Arm/Group | P07535 Study Participants With a TOF Ratio <0.9 | P07535 Study Participants With a TOF Ratio ≥0.9
Number analyzed (Participants) | 64 | 193
participants
  Participants Receiving Propofol | 60 | 169
  Participants Receiving Sevoflurane | 4 | 24

4. Secondary Outcome: Number of Participants With and Without Postoperative Residual Neuromuscular Blockade Who Received Neuromuscular Blockade Reversal Agents
Description: Neuromuscular blockade reversal agents administered to participants undergoing surgical procedures were recorded. The number of participants who received such an agent is presented, for participants with and without residual neuromuscular blockade.
Time Frame: From end of surgery through PACU arrival, an expected average of 10 minutes
Population: FAS population includes all treated participants
Measure: Number; unit: participants
Arm/Group | P07535 Study Participants With a TOF Ratio <0.9 | P07535 Study Participants With a TOF Ratio ≥0.9
Number analyzed (Participants) | 91 | 259
participants | 71 | 162
Statistical Analysis 1: Comparison: P07535 Study Participants With a TOF Ratio <0.9 vs P07535 Study Participants With a TOF Ratio ≥0.9; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.01, Chi-square test or Fisher's Exact Test

5. Secondary Outcome: Number of Participants With and Without Postoperative Residual Neuromuscular Blockade With Postoperative Events
Time Frame: From end of surgery through hospital discharge, an expected average of 6 days
Population: FAS population includes all treated participants
Measure: Number; unit: participants
Arm/Group | P07535 Study Participants With a TOF Ratio <0.9 | P07535 Study Participants With a TOF Ratio ≥0.9
Number analyzed (Participants) | 91 | 259
participants | 12 | 21

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 3/350
Other Adverse Events (participants affected / at risk) | 0/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=350)
respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
septic shock (Infections and infestations) | 1 (1)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may not publish/publicly present interim results without prior consent of Sponsor. Any materials that report results of the study must be sent to Sponsor 45 days prior to submission for publication/presentation. Sponsor has right to review and comment. In case of any disagreements concerning appropriateness of the materials, investigator and Sponsor must meet to make a good faith effort to discuss/resolve the issues or disagreement, prior to submission for publication/presentation.